CLINICAL TRIAL: NCT01927380
Title: Autonomic Nervous System Modulation During Laparoscopic Prostatectomy
Status: Completed | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, MD, ASST Fatebenefratelli Sacco
Other Study IDs: CE#371/2013
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Intervention Affecting Autonomic Nervous System
Keywords: autonomic nervous system modulation; heart rate variability; prostatectomy; steep trendelenburg; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- brachytherapy: males undergoing elective laparoscopic radical prostatectomy steep trendelenburg position with pneumoperitoneum
  Interventions: Other: steep trendelenburg position with pneumoperitoneum

INTERVENTIONS:
Other: steep trendelenburg position with pneumoperitoneum — ANS activity and baroreflex modulation is assessed at (i) baseline; (ii) after induction of general anesthesia; (iii) after steep trendelenburg position (head down at 25 degrees); (iv) after induction of pneumoperitoneum and (v) after removal of trendelenburg and pneumoperitoneum

SUMMARY:
The purpose of this study is to measure the variations of autonomic nervous system (ANS) modulation directed to the heart and vessels induced by pneumoperitoneum and steep trendelenburg position.

DETAILED DESCRIPTION:
The association of pneumoperitoneum and steep trendelenburg position, commonly used during laparoscopic radical prostatectomy, leads to significant changes in hemodynamics. Many studies found modifications of cardiac output, stroke work index, arterial pressure, central vein pressure and wedge pressure. Moreover, there are reports of severe bradycardia and cardiac arrest following pneumoperitoneum in association with steep trendelenburg. A vagal hypertone (induced by the combination of these two factors) or sympathetic hypractivity (elicited by pneumoperitoneum) had been alternatively postulated to cause these hemodynamic changes. To date there are not sufficient physiologic evidences of modification of ANS activity during steep trendelenburg position in association with pneumoperitoneum.

ANS modulation is studied non invasively by means of heart rate variability and baroreflex sensitivity. Beat-to-beat intervals are computed detecting the QRS complex on the ECG and locating the R-apex using parabolic interpolation. The maximum arterial pressure within each R-to-R interval is taken as systolic arterial pressure (SAP). Sequences of 300 values are randomly selected inside each experimental condition. The power spectrum is estimated according to a univariate parametric approach fitting the series to an autoregressive model. Autoregressive spectral density is factorized into components each of them characterized by a central frequency. A spectral component is labeled as LF if its central frequency is between 0.04 and 0.15 Hz, while it is classified as HF if its central frequency is between 0.15 and 0.4 Hz. The HF power of R-to-R series is utilized as a marker of vagal modulation directed to the heart , while the LF power of SAP series is utilized as a marker of sympathetic modulation directed to vessels. The ratio of the LF power to the HF power assessed from R-to-R series is taken as an indicator simpatho-vagal balance directed to the heart. Baroreflex control in the low frequencies is computed as the square root of the ratio of LF(RR) to LF(SAP). Similarly baroreflex control in the high frequencies is defined as the square root of the ratio of HF(RR) to HF(SAP).

The optic nerve sheet's diameter is assessed echographically after induction of general anesthesia and at the end of the surgery.

Management of general anesthesia is standardized:

* induction with propofol 1.5-2 mg/kg, Remifentanil Target Controlled Infusion (TCI) Ce 4 ng/ml , neuromuscolar blockade with cisatracurium 0.2 mg/kg.
* Maintenance: Sevoflurane 0.6-1.5 MAC (State Entropy target: 40-60); Remifentanil TCI (range Ce 3-15 ng/ml) (Surgical Pleth Index target: 20-50).
* mechanical ventilation at respiratory rate ≥14 breats/min, with tidal volume adjusted to maintain end-tidal carbon dioxide at 32-38 mmHg, and Pplateu <32 cmH2O.

Sample size:

to detect a difference in LF/HF ratio of 0.8 with a SD of 1.7, a power of 0.80 and type I error of 0.05, 37 patients are needed.

ELIGIBILITY:
Inclusion Criteria:

* males scheduled for elective laparoscopic prostatectomy
* sinus rhythm at ECG
* ectopic heart beats <5% of all heart beats
* american society of anesthesiologists status 1-3

Exclusion Criteria:

* autonomic dysfunction (documented or suspected)
* adrenal or thyroid dysfunction
* organ dysfunction secondary to diabetes (i.e. nephropathy, retinopathy, neuropathy)
* history of stroke, traumatic spinal injury, heart surgery or major vascular surgery
* intracranial hypertension (documented or suspected)
* hydrocephalus
* cardiac functional status ≥NYHA IIb
* non sinusal heart rhythm
* ectopic heart beats ≥5% of normal heart beats
* therapy with beta-blockers or beta2-agonists

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human males undergoing elective laparoscopic prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To measure the changes of ANS modulation directed to the heart and to the vessels, and the changes of baroreflex control induced by steep trendelenburg position and pneumoperitoneum | Day of surgery

SECONDARY OUTCOMES:
To measure the correlation between ANS changes and hemodynamics | day of surgery

OTHER OUTCOMES:
to measure changes of the optic nerve sheet's diameter during steep trendelenburg and pneumoperitoneum | day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinando Raimondi, Director, Study Chair — Azienda Ospedaliera "L.Sacco"; Riccardo Colombo, Consultant, Principal Investigator — Azienda Ospedaliera "L.Sacco"; Stefano Guzzetti, Director, Study Director — Azienda Ospedaliera "L.Sacco"
Locations (1):
- Azienda Ospedaliera "Luigi Sacco" - Polo Universitario - University of Milan, Milan, Italy

REFERENCES:
- [Background] Falabella A, Moore-Jeffries E, Sullivan MJ, Nelson R, Lew M. Cardiac function during steep Trendelenburg position and CO2 pneumoperitoneum for robotic-assisted prostatectomy: a trans-oesophageal Doppler probe study. Int J Med Robot. 2007 Dec;3(4):312-5. doi: 10.1002/rcs.165. PMID 18200624
- [Background] Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol. 2009 May;55(5):1037-63. doi: 10.1016/j.eururo.2009.01.036. Epub 2009 Jan 25. PMID 19185977
- [Background] Park EY, Koo BN, Min KT, Nam SH. The effect of pneumoperitoneum in the steep Trendelenburg position on cerebral oxygenation. Acta Anaesthesiol Scand. 2009 Aug;53(7):895-9. doi: 10.1111/j.1399-6576.2009.01991.x. Epub 2009 May 6. PMID 19426238
- [Background] Awad H, Santilli S, Ohr M, Roth A, Yan W, Fernandez S, Roth S, Patel V. The effects of steep trendelenburg positioning on intraocular pressure during robotic radical prostatectomy. Anesth Analg. 2009 Aug;109(2):473-8. doi: 10.1213/ane.0b013e3181a9098f. PMID 19608821
- [Background] Amini A, Kariman H, Arhami Dolatabadi A, Hatamabadi HR, Derakhshanfar H, Mansouri B, Safari S, Eqtesadi R. Use of the sonographic diameter of optic nerve sheath to estimate intracranial pressure. Am J Emerg Med. 2013 Jan;31(1):236-9. doi: 10.1016/j.ajem.2012.06.025. Epub 2012 Aug 31. PMID 22944553
- [Background] Lestar M, Gunnarsson L, Lagerstrand L, Wiklund P, Odeberg-Wernerman S. Hemodynamic perturbations during robot-assisted laparoscopic radical prostatectomy in 45 degrees Trendelenburg position. Anesth Analg. 2011 Nov;113(5):1069-75. doi: 10.1213/ANE.0b013e3182075d1f. Epub 2011 Jan 13. PMID 21233502
- [Background] Haas S, Haese A, Goetz AE, Kubitz JC. Haemodynamics and cardiac function during robotic-assisted laparoscopic prostatectomy in steep Trendelenburg position. Int J Med Robot. 2011 Dec;7(4):408-13. doi: 10.1002/rcs.410. Epub 2011 Aug 3. PMID 21815239
- [Background] Crystal GJ, Salem MR. The Bainbridge and the "reverse" Bainbridge reflexes: history, physiology, and clinical relevance. Anesth Analg. 2012 Mar;114(3):520-32. doi: 10.1213/ANE.0b013e3182312e21. Epub 2011 Sep 29. PMID 21965361
- [Background] Montano N, Ruscone TG, Porta A, Lombardi F, Pagani M, Malliani A. Power spectrum analysis of heart rate variability to assess the changes in sympathovagal balance during graded orthostatic tilt. Circulation. 1994 Oct;90(4):1826-31. doi: 10.1161/01.cir.90.4.1826. PMID 7923668
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Pagani M, Montano N, Porta A, Malliani A, Abboud FM, Birkett C, Somers VK. Relationship between spectral components of cardiovascular variabilities and direct measures of muscle sympathetic nerve activity in humans. Circulation. 1997 Mar 18;95(6):1441-8. doi: 10.1161/01.cir.95.6.1441. PMID 9118511
- [Background] Ray CA. Interaction of the vestibular system and baroreflexes on sympathetic nerve activity in humans. Am J Physiol Heart Circ Physiol. 2000 Nov;279(5):H2399-404. doi: 10.1152/ajpheart.2000.279.5.H2399. PMID 11045977
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Derived] Colombo R, Agarossi A, Borghi B, Ottolina D, Bergomi P, Ballone E, Minari C, Della Porta V, Menozzi E, Figini S, Fossali T, Catena E. The effect of prolonged steep head-down laparoscopy on the optical nerve sheath diameter. J Clin Monit Comput. 2020 Dec;34(6):1295-1302. doi: 10.1007/s10877-019-00418-5. Epub 2019 Nov 5. PMID 31691148